CLINICAL TRIAL: NCT07095686
Title: An Open-Label Study of an Experimental Antisense Oligonucleotide Treatment for Amyotrophic Lateral Sclerosis (ALS) Due to an Arg15Leu Pathogenic Variant in CHCHD10
Brief Title: Personalized Antisense Oligonucleotide for Participants With CHCHD10 ALS
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV3923
Record Dates: First submitted 2025-05-12; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label nL-CHCHD-001 (Experimental)
  Interventions: Drug: nL-CHCHD-001

INTERVENTIONS:
Drug: nL-CHCHD-001 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for individual participants with amyotrophic lateral sclerosis (ALS) due to a pathogenic variant in CHCHD10

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representatives(s)
* Ability to travel to the study site and adhere to study related follow-up examinations and/or procedures and provide access to participant's medical records
* Genetically confirmed neurological disorder

Exclusion Criteria:

* Participant has any condition that in the opinion of the Site Investigator would ultimately prevent the completion of study procedures
* Use of an investigational medication within less than 5 half-lives of the drug at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R).
Motor Function | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in Slow Vital Capacity (SVC)
Motor Function | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in muscle strength as quantified by Handheld Dynamometry (HHD)
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in Edinburgh Cognitive and Behavioral ALS Screen (ECAS) score
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on ALS Cognitive Behavioral Screen (ALS-CBS)
Clinical Functioning | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in scores on Amyotrophic Lateral Sclerosis Assessment Questionnaire 5 (ALSAQ-5)

SECONDARY OUTCOMES:
Disease Biomarkers | Baseline to 12 months
  Change from baseline at 12-months post nL-CHCHD-001 administration in serum and CSF neurofilament light chain levels
Safety and Tolerability | Baseline to 12 months
  Incidence and severity of Adverse Events
Safety and tolerability | Baseline to 12 months
  Emergent abnormalities in physical exam (changes in appearance, skin, neck, ears, nose, throat, heart/lungs, abdomen, lymph nodes, and extremities compared to baseline)
Safety and Tolerability | Baseline to 12 months
  Emergent abnormalities in neurological exam (changes in mental status, gait, cerebellar, cranial nerve, motor, reflex, and sensations compared to baseline)
Safety and tolerability | Baseline to 12 months
  Emergent abnormalities in laboratory analyses (results outside of normal range for CSF, chemistry, hematology, coagulation, and urinalysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, Irving Medical Center, New York, New York, United States